CLINICAL TRIAL: NCT01701596
Title: Safety and Efficacy of Immediate Rotational Atherectomy in Nondilatable Calcified Lesion Complicated by Coronary Dissection (RAISE)
Brief Title: Safety and Efficacy of Rotational Atherectomy (RA) in Coronary Dissection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAISE
Record Dates: First submitted 2012-09-28; First posted 2012-10-05 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Artery Disease
Keywords: Rotational atherectomy; Coronary dissection; Percutaneous coronary intervention; Calcification
MeSH Terms: conditions — Coronary Artery Disease; Calcinosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rotational atherectomy (RA) (Experimental): Immediate rotational atherectomy (RA) in the treatment with nondilatable calcified lesion complicated by coronary dissection
  Interventions: Procedure: Immediate rotational atherectomy (RA)
- Delayed rotational atherectomy (RA) (Active Comparator): Delayed RA in the treatment with nondilatable calcified lesion complicated by coronary dissection
  Interventions: Procedure: Delayed rotational atherectomy (RA)

INTERVENTIONS:
Procedure: Immediate rotational atherectomy (RA) — Immediate RA in the treatment with nondilatable calcified lesion complicated by coronary dissection.
  Arms: Rotational atherectomy (RA)
Procedure: Delayed rotational atherectomy (RA) — Delayed RA in the treatment with nondilatable calcified lesion complicated by coronary dissection
  Arms: Delayed rotational atherectomy (RA)

SUMMARY:
This study is aimed at examining the safety and efficacy of rotational atherectomy (RA) in nondilatable calcified lesion complicated by coronary dissection during percutaneous coronary intervention (PCI) procedure.

DETAILED DESCRIPTION:
Coronary artery dissection is a contraindication for the use of rotational atherectomy, since rotational atherectomy may propagate coronary dissection. In the presence of coronary dissection, conservative management is suggested for approximately 4 weeks to permit the dissection to heal prior to treatment with rotational atherectomy. However, a lot of patients have frequent angina attacks and some patients develop serious complications including abrupt vessel closure during this period. Thus, immediate strategies cope with coronary dissection induced by balloon dilation is needed for the early recovery of those patients. The present study was performed to compare the safety and efficacy of immediate RA and delayed RA in the treatment with nondilatable calcified lesion complicated by coronary dissection.

ELIGIBILITY:
Inclusion Criteria:

* age between 30 and 85 years old
* nondilatable calcified lesion complicated by coronary dissection during percutaneous coronary intervention (PCI) procedure
* Coronary artery dissection type A, B and type C according to the National Heart, Lung and Blood Institute (NHLBI) coronary dissection criteria

Exclusion Criteria:

* acute myocardial infarction
* unprotected left main stenosis
* chronic total occlusion
* saphenous vein graft lesion
* cardiomyopathy
* severe valvular heart disease
* NYHA functional class IV heart failure at baseline
* chronic renal failure on hemodialysis
* severe lung and liver disease or cancer

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2004-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
All cause death | 4 years
  cardiac death and non-cardiac death

SECONDARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | 4 years
6-min walk distance (6MWD) | 4 years
angina class | 4 years
  angina class according to the Canadian Cardiovascular Society (CCS) classification and Seattle Angina Questionnaire
Non-fatal myocardial infarction | 4 years
Stent thrombosis | 4 years
Cardiac tamponade | 4 years
Stroke | 4 years
Target lesion revascularization | 4 years
New York Heart Association (NYHA) class IV heart failure | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Chengxiang Li, M.D., Ph.D., Principal Investigator — Department of Cardiolody, Xijing Hospital, Fourth Military Medical University
Locations (1):
- Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China